CLINICAL TRIAL: NCT02082860
Title: Phase I, Multicentre, Open Label, Single Dose, Dose-ranging Clinical Trial to Investigate the Safety and Tolerability of a Gene Therapy rAAV2/5-PBGD for the Treatment of Acute Intermittent Porphyria
Brief Title: Phase I Gene Therapy Clinical Trial Using the Vector rAAV2/5-PBGD for the Treatment of Acute Intermittent Porphyria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Digna Biotech S.L. (Industry)
Collaborators: Porphyria Centre Sweden (Unknown); University of Navarra (Other); UniQure N.V. (Industry); Nationales Centrum für Tumorerkrankungen (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAVPBGD-AIP-001; 2011-005590-23 (EudraCT Number)
Record Dates: First submitted 2014-02-28; First posted 2014-03-10 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Acute Intermittent Porphyria
Keywords: Porphyria; Gene therapy; AAV; Liver gene transfer
MeSH Terms: conditions — Porphyria, Acute Intermittent; Porphyrias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort A (Experimental): rAAV2/5-PBGD vector dosage 1
  Interventions: Genetic: rAAV2/5-PBGD vector dosage 1
- Cohort B (Experimental): rAAV2/5-PBGD vector dosage 2
  Interventions: Genetic: rAAV2/5-PBGD vector dosage 2
- Cohort C (Experimental): rAAV2/5-PBGD vector dosage 3
  Interventions: Genetic: rAAV2/5-PBGD vector dosage 3
- Cohort D (Experimental): rAAV2/5-PBGD vector dosage 4
  Interventions: Genetic: rAAV2/5-PBGD vector dosage 4

INTERVENTIONS:
Genetic: rAAV2/5-PBGD vector dosage 1 — Intravenous injection of rAAV2/5-PBGD vector, single administration on Day 1.
  Arms: Cohort A
Genetic: rAAV2/5-PBGD vector dosage 2 — Intravenous injection of rAAV2/5-PBGD vector, single administration on Day 1.
  Arms: Cohort B
Genetic: rAAV2/5-PBGD vector dosage 3 — Intravenous injection of rAAV2/5-PBGD vector, single administration on Day 1.
  Arms: Cohort C
Genetic: rAAV2/5-PBGD vector dosage 4 — Intravenous injection of rAAV2/5-PBGD vector, single administration on Day 1.
  Arms: Cohort D

SUMMARY:
This is a Phase I trial aimed to determine the safety of the investigational gene therapy product (rAAV2/5-PBGD) for the treatment of Acute Intermittent Porphyria (AIP).

Up to eight patients fulfilling the eligibility criteria will participate in this multicentre, open label, single dose, dose-ranging Phase I clinical trial.

The enrolled patients will be followed up to assess the safety profile of the investigational gene therapy product and to establish the maximum therapeutic safe dose to be administered in future confirmatory/pivotal clinical trial(s). In addition, the biological and clinical response to the treatment with rAAV2/5-PBGD in AIP patients will be assessed.

A complete evaluation of the clinical (symptoms and quality of life assessment) and laboratory (blood and urine) data will be performed.

DETAILED DESCRIPTION:
Acute Intermittent Porphyria (AIP) is inherited as an autosomal dominant disorder of the heme biosynthesis pathway. AIP is caused by a genetic defect in porphobilinogen deaminase (PBGD), a key enzyme for heme synthesis.

AIP is characterized by acute episodes and asymptomatic periods. Neuropathic symptoms are predominantly in these attacks, which may be related to the toxic effect produced by the precursors delta-aminolevulinic acid (ALA) and porphobilinogen (PBG), accumulated because the enzyme deficiency. It occurs with very low prevalence (1 in 50,000), but figures for prevalence based on clinical manifestations (i.e., acute attacks) greatly underestimate the number of patients with latent AIP.

Abdominal pain is the most common symptom, sometimes with constipation. Paresthesia and paralysis also occur, and death may result from respiratory paralysis. Other symptoms, including seizures, psychotic episodes, and hypertension, develop during acute attacks. They may be precipitated by porphyrogenic drugs such as barbiturates, progestogens and sulfonamides, some of which are known to induce the first rate-controlling step in heme synthesis, ALA synthesis. Other known precipitants are alcohol, infection, starvation, and hormonal changes; attacks are more common in women. Acute attacks rarely occur before puberty.

This is a Phase I clinical trial mainly aimed to evaluate the safety of a recombinant adeno associated vector with a liver-specific promoter for the PBGD expression (rAAV2/5-PBGD), for the treatment of Acute Intermittent Porphyria.

The patients will be enrolled in an adaptive dose-escalation, multicentre trial to assess safety profile, and to establish the maximum therapeutic safe dose to be administrated to patients in further confirmatory or pivotal clinical trial.

This clinical trial is preceded by an "Observational study of acute intermittent porphyria patients" (DIG-API-2011-01). In this observational study, severe AIP patients have been followed for 6 to up to a maximum 24 months. During this time, the clinical and laboratory (blood and urine biochemistry) conditions of the patients were evaluated, in order establish clinical and biological baseline and history to compare the future results of this clinical trial.

During this clinical trial, the safety will be evaluated by the Adverse Events (AEs) and Serious Adverse Events (SAEs) assessment. A complete evaluation of the clinical and laboratory (blood and urine) data will be collected. The study will also investigate as secondary endpoints the effect of this treatment to modify other aspects of the patient condition.

Due to the heterogeneity of genetic mutations and inter-individual variation, clinical symptomatology and ALA/PBG levels in AIP subjects showed an evident variability in urine samples both during acute attacks and during remission; each subject will be its own control, so this study will be an intra-individually controlled clinical trial. At the end of the clinical trial the efficacy evaluation will be performed based on the clinical and biochemical changes compared to the baseline established in the previous observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patient's written Informed Consent
* Age between 18 and 64 years, inclusively.
* Patients with confirmed diagnosis of Acute Intermittent Porphyria(AIP), as confirmed by clinical, biochemical data and genetic confirmation of porphobilinogen deaminase (PBGD) gene mutation. The patient must have a severe AIP condition, with at least two hospitalizations during the previous year due to acute attacks (clinical manifestations of acute porphyria), or at least four hospitalizations during the previous year due to the requirement of hospital treatment administration (including day-hospital and home hospital program)
* Previous participation in the "Observational study of acute intermittent porphyria patients" for at least six months.
* Ability to follow instructions and cooperate during the study conduct

Exclusion Criteria:

* Pregnant women, as confirmed by a positive urine pregnancy test, or with intention of becoming pregnant
* Female subjects of childbearing potential who are not using barrier methods of contraception, at least during the study.
* Male subjects with partners of child bearing potential who are not using barrier contraceptive methods, at least during the study
* Acute or chronic liver disease of viral, autoimmune or metabolic causes
* History of acute or chronic severe gastrointestinal dysfunction (different than those typical gastrointestinal symptoms associated with an acute attack of AIP), in the opinion of the principal investigator
* Kidney disorder (renal impairment defined as plasma creatinine > 2 mg/dl (150 µmol/l)), severe respiratory disease, severe autoimmune disease or severe acute active infection
* Evidence of active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection as reflected by HBs antigen or HCV-antibodies positivity (in case of HCV-antibodies positivity a HCV-RNA test should be performed in order to confirm active viral replication)
* Positive human immunodeficiency virus (HIV) serological test
* History of drug use (cannabis, cocaine, amphetamines, barbiturates) or alcohol abuse or addiction, during the three months preceding the selection visit
* Presence of neutralizing antibodies against adeno-associated serotype 5 (AAV5)
* Current or previous (within the previous 12 months) participation in a gene therapy trial.
* Previous participation (at any time) in a gene therapy trial using AAV vectors
* Any other disease or condition that, in the opinion of the principal investigator, contraindicates the participation in the study because it can expose the patient to a risk or because it disqualifies the patient to complete the schedule of the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with Adverse Events and Serious Adverse Events | Up to 48 weeks
  To assess the safety and determine the maximum therapeutic safe dose of the investigational gene therapy (GT) product rAAV2/5-PBGD for the treatment of AIP, registering and evaluating the occurrence of Adverse Events and/or Serious Adverse Events at the dose identified will be performed

SECONDARY OUTCOMES:
Effect of the treatment on porphobilinogen (PBG) and delta-aminolevulinic acid (ALA) urinary level. | Up to 48 weeks
Clinical evolution of acute intermittent porphyria. Frequency of hospitalizations | Up to 48 weeks
Frequency of treatments for AIP symptoms | Up to 48 weeks
  The information regarding the requirement of specific treatments for symptoms control (analgesics, hemin and glucose endovenous solutions) will be collected.
Psychological evaluation of AIP patients | Up to 48 weeks
  Anxiety and depression will be assessed by using the Beck Anxiety Inventory (BAI) and Beck Depression Inventory (BDI) rating scales.
Health related quality of life of AIP patients | Up to 48 weeks
  Health-related quality of life will be assessed through the SF-36v2 questionnaire
Frequency of AIP symptoms | Up to 48 weeks
Pharmacokinetic parameters | Selection visit, Days 1, 2 and 3, week 1, week 2, week 3 and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ruiz, MD, Study Chair — Digna Biotech S.L.; Jesus Prieto, MD, Principal Investigator — Clinica Universidad de Navarra; Rafael Enriquez de Salamanca, MD, Principal Investigator — Hospital 12 de Octubre
Locations (2):
- Spain (2):
  - 12 Octubre Hospital, Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre

REFERENCES:
- [Derived] D'Avola D, Lopez-Franco E, Sangro B, Paneda A, Grossios N, Gil-Farina I, Benito A, Twisk J, Paz M, Ruiz J, Schmidt M, Petry H, Harper P, de Salamanca RE, Fontanellas A, Prieto J, Gonzalez-Aseguinolaza G. Phase I open label liver-directed gene therapy clinical trial for acute intermittent porphyria. J Hepatol. 2016 Oct;65(4):776-783. doi: 10.1016/j.jhep.2016.05.012. Epub 2016 May 17. PMID 27212246